CLINICAL TRIAL: NCT06935851
Title: The Effect of Word Characteristics and Orthography on Vocabulary Learning
Brief Title: Effect of Word Characteristics and Orthography on Vocabulary Learning
Acronym: VOCAL+
Status: Active, not recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: Mariana Silva (Other)
Collaborators: Arizona State University (Other)
Responsible Party: Sponsor-Investigator, Mariana Silva, Doctoral Student, Arizona State University
Organization: Arizona State University (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: STUDY00020728
Record Dates: First submitted 2024-12-17; First posted 2025-04-20 (Actual); Last update posted 2025-04-20 (Actual); Status verified 2025-04

CONDITIONS: Developmental Child Delay

STUDY DESIGN:
Intervention Model Description: Single group assignment
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Single group Assignment (Other): There are no subgroups in this study. All participants will receive the intervention.
  Interventions: Behavioral: VOCAB +

INTERVENTIONS:
Behavioral: VOCAB + — The purpose of the study is to investigate how word characteristics (e.g., phonotactic probability) and orthography effect vocabulary learning by children with low oral language levels. We will be using a 2 x 2 within-subjects factorial design where every participant serves as their own control. This 12-week study aims to improve the Efficiency of vocabulary learning for children with low oral language levels.
  The four interventions that are all participants will be exposed to are the following: high pp words with orthography; high pp words without orthography; low pp words with orthography; low pp words without orthography.

SUMMARY:
The purpose of the study is to investigate how word characteristics (e.g., phonotactic probability) and orthography affect vocabulary by children with low oral language levels. The investigators will use a 2 x 2 within-subjects factorial design where every participant receives the treatment. This 12-week study aims to improve vocabulary learning efficiency for children with low oral language levels. The study's findings will uniquely contribute to the field in that this is the first research study using real words instead of nonwords while combining word learning research with vocabulary learning.

DETAILED DESCRIPTION:
The investigators are proposing a vocabulary intervention that analyzes word sounds and sound segments. This analysis offers valuable insights into how children at risk for specific learning disabilities, such as dyslexia or speech and language impairments, learn words differently from typically developing children.

ELIGIBILITY:
Inclusion Criteria:

Score of 85 or lower on the Clinical Evaluation of Language Fundamentals - CELF (4) Enrolled in or just completed third grade.

Exclusion Criteria:

Any diagnosis of sensory impairments A diagnosis of autism or traumatic brain injury

Ages: 8 Years to 9 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 23 (Actual)
Dates: Start 2025-02-03 (Actual); Primary Completion 2025-04-25 (Estimated); Study Completion 2025-05-21 (Estimated)

PRIMARY OUTCOMES:
Pre- and post test total correct scores | up to 12 weeks
  Is there a significant difference in pre- and post test total correct scores for different word types with mother's education level covaried as measured by comprehension, recognition, production, spelling recognition and spelling production.

SECONDARY OUTCOMES:
Number of trials to criterion | up to 8 weeks
  Is there a significant difference in the number of trials to criterion required to learn a new word for different word types as measured by comprehension, recognition, production, spelling recognition and spelling production?

OTHER OUTCOMES:
Total number of words learned to criterion | 12 weeks
  Is there a significant difference in the total number of words learned to criterion comprehension, recognition, production, spelling recognition, and spelling production?

CONTACTS AND LOCATIONS:
Locations (1):
- Osborn District School Encanto, Phoenix, Arizona, United States

IPD SHARING:
Plan to Share IPD: Yes
* Study Protocol
  * Statistical Analysis Plan (SAP)
  * Informed Consent Form
  * Clinical Study Report
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: The data will be made available within 7 months of the study's conclusion and will remain available for at least 5 years.
Access Criteria: Signing a data use agreement.
URL: https://osf.io

REFERENCES:
- Available data/document: Study Protocol — https://osf.io — signing a data agreement

DOCUMENTS (1):
  • Statistical Analysis Plan (2024-12-17): https://cdn.clinicaltrials.gov/large-docs/51/NCT06935851/SAP_000.pdf